CLINICAL TRIAL: NCT06884254
Title: A Phase 3, Randomized, Multicenter, Parallel-arm, Double-blind Study to Compare Efficacy and Safety of EG1206A (EirGenix' Pertuzumab) and Perjeta® (Pertuzumab) Sourced From EU as Neoadjuvant Treatment in Combination With Trastuzumab and Chemotherapy in Patients With HER2-positive Hormone Receptor-negative Early Breast Cancer
Brief Title: Efficacy and Safety Study of EG1206A (EirGenix' Pertuzumab) Compared With EU-sourced Perjeta® (Pertuzumab) in Patients With HER2-positive Hormone Receptor Negative Early Breast Cancer.
Acronym: EGC102
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Following SA from both the US FDA and the EMA, EirGenix, Inc. has decided to streamline the clinical-development program for EG1206A (biosimilar to Perjeta). EirGenix has concluded that the continuation of the study in no longer necessary.
Sponsor: EirGenix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EGC102; 2024-518619-21-00 (EU CTIS Number)
Record Dates: First submitted 2025-03-18; First posted 2025-03-19 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Early Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pertuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- EG1206A (Experimental): During the neoadjuvant treatment period, patients will receive 6 cycles with EG1206A, trastuzumab, and chemotherapy (docetaxel and carboplatin), followed by surgery.
  If criteria to remain on study are still fulfilled, patients will continue treatment in the adjuvant setting, starting 2 to 6 weeks after surgery. Patients will receive 12 cycles with EG1206A and trastuzumab (as originally randomized in the neoadjuvant part) to complete 1 year of HER2-targeted therapy.
  Interventions: Drug: EG1206A
- Perjeta (Active Comparator): During the neoadjuvant treatment period, patients will receive 6 cycles with Perjeta, trastuzumab, and chemotherapy (docetaxel and carboplatin), followed by surgery.
  If criteria to remain on study are still fulfilled, patients will continue treatment in the adjuvant setting, starting 2 to 6 weeks after surgery. Patients will receive 12 cycles with Perjeta and trastuzumab (as originally randomized in the neoadjuvant part) to complete 1 year of HER2-targeted therapy.
  Interventions: Drug: Perjeta

INTERVENTIONS:
Drug: EG1206A — EG1206A 420mg is ongoing to be administered after 840mg loading dose.
  Arms: EG1206A
Drug: Perjeta — Perjeta 420mg is ongoing to be administered after 840mg loading dose.
  Arms: Perjeta

SUMMARY:
The purpose of this research study is to compare the efficacy and safety of EG1206A with Perjeta in combination with trastuzumab and chemotherapy as neoadjuvant treatment for 18 weeks, followed by surgery and subsequent EG1206A or Perjeta in combination with trastuzumab, as adjuvant treatment for 36 weeks.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (before randomization)

Patients are eligible to be included in the study only if all of the following criteria apply:

1. Provide signed and dated written informed consent before any study related procedures are performed. The informed consent will cover both parts of the study (neoadjuvant part and adjuvant part).
2. Female and male patients ≥ 18 and ≤ 70 years of age.
3. Histologically-confirmed invasive carcinoma of the breast.
4. Early stage (T2-3, N0-1, M0), locally advanced stage (T2-3, N2-3, M0 or T4a-c, any N, M0), or inflammatory (T4d, any N, M0) breast cancer planned for surgical resection (mastectomy or lumpectomy of the breast, and resection of sentinel or axillary lymph nodes).
5. Unilateral, measurable tumor of the breast > 2 cm in diameter (by ultrasound and/or mammography).
6. HER2-positive tumor status (according to American Society of Clinical Oncology/College of American Pathologists [ASCO/CAP] guidelines [2018, 2023]), as confirmed by central laboratory.
7. Estrogen receptor and progesterone receptor-negative tumor (according to ASCO/CAP guidelines [2020]), as confirmed by central laboratory.
8. Eastern Cooperative Oncology Group (ECOG) score of 0 or 1.
9. Baseline left ventricular ejection fraction (LVEF) ≥ 55%, measured by echocardiography or MUGA (multigated acquisition scan).
10. Adequate bone marrow function, defined as neutrophil count of ≥ 1,500/µL, hemoglobin ≥ 9 g/dL, and platelet count of ≥ 100,000/µL.
11. Adequate hepatic and renal function, defined as total bilirubin ≤ 1.5 × upper limit of normal (ULN) (or ≤ 3 × ULN and direct bilirubin within normal limits in patients with well documented Gilbert's syndrome), alanine aminotransferase (ALT) ≤ 3 × ULN, aspartate aminotransferase (AST) ≤ 3 × ULN, creatinine clearance ≥ 30 mL/min (according to Cockcroft and Gault equation).
12. International normalized ratio ≤ 1.5 × ULN (2 to 3 × ULN if on anticoagulants with vitamin K antagonists) or prothrombin time ≤ 1.5 × ULN; activated partial thromboplastin time ≤ 1.5 × ULN.
13. For women of childbearing potential (WOCBP): WOCBP must have a negative serum pregnancy test at Screening and must use adequate birth control. Adequate birth control is defined as agreement to consistently practice an effective and accepted method of contraception throughout the duration of the study and for 7 months after the End of Treatment (EOT) Visit. These methods include hormonal contraceptives, intrauterine device, or double barrier contraception (i.e., condom + diaphragm) or a male partner with documented vasectomy. Non-childbearing potential is defined as post-menopausal for at least 1 year or surgical sterilization or hysterectomy at least 3 months before study start. Women will be considered post-menopausal if they have been amenorrheic for 12 months without an alternative medical cause.
14. For men: Men must agree to use reliable contraceptive measures throughout the duration of the study and for 7 months after the EOT Visit. These methods include documented vasectomy, double-barrier contraception (i.e., condom and diaphragm), or true sexual abstinence (when this is in line with the preferred and usual lifestyle of the patient).

    Inclusion Criteria (after surgery for the adjuvant part of the study)
15. Patients with complete pathological remission.
16. Patients with residual disease that cannot receive further treatment with trastuzumab emtansine (in case of contraindication to trastuzumab emtansine, recommendations from local guidelines, or at the discretion of the Investigator).

Exclusion Criteria:

1. Stage IV (metastatic) breast cancer, bilateral breast cancer.
2. Pregnancy or lactation or considering becoming pregnant.
3. Previous treatment (chemotherapy, biologic therapy, radiation, or surgery) for invasive malignant disease or other concomitant malignancy, other than basal cell carcinoma of the skin. Previous treatment for carcinoma in situ of the cervix is allowed.
4. Previous treatment with Perjeta.
5. Active hepatitis B or hepatitis C infection, or infection with the human immunodeficiency virus (HIV) as shown by a positive diagnostic test for hepatitis B virus (HBV), hepatitis C virus (HCV) or HIV.
6. History of or existing congestive heart failure (CHF) New York Heart Association class II or higher; angina pectoris or arrhythmia requiring medication; poorly controlled hypertension; history of myocardial infarction or cardiac failure; clinically significant cardiac valvular disease; hemodynamic effective pericardial effusion; other cardiomyopathies.
7. Any investigational treatment less than 30 days prior to study entry, or within a time interval less than at least 5 half-lives of the investigational medicinal product (IMP: EG1206A or Perjeta), whichever is longer.
8. Hypersensitivity to the IMP (EG1206A or Perjeta), trastuzumab or trastuzumab biosimilar, carboplatin (or other platin compounds), and docetaxel, or to any of their excipients.
9. Vaccination with live attenuated vaccines during the study.
10. History of, or known current problems with, drug or alcohol abuse.
11. Other serious illness, previous surgery (other than for invasive malignant disease), medical disorder or condition that, in the opinion of the Investigator, would make the patient unsuitable for participation in the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-05 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Determination of pathologic complete response (pCR) at time of surgery | At the time of surgery (3-6 weeks after completion of neoadjuvant chemotherapy)
  • pCR at time of surgery, where pCR is defined as the absence of residual invasive cancer of the complete resected breast specimen (regardless of ductal carcinoma in situ [DCIS]) and all sampled sentinel and/or axillary lymph nodes (ypT0/is ypN0), as assessed by central laboratory.

CONTACTS AND LOCATIONS:
Locations (1):
- Methodist Health System Clinical Research Institute, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided